CLINICAL TRIAL: NCT04102072
Title: The Consistency of Cardiac Output Measurements by Different Methods in VA-ECMO Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COMMENT
Record Dates: First submitted 2019-09-10; First posted 2019-09-25 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Extracorporeal Membrane Oxygenation
Keywords: pulmonary artery catheter; echocardiography; fluid responsiveness; extracorporeal membrane oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trendelenburg Maneuver (Experimental): The Trendelenburg position is a common treatment in medicine.It is used either as a diagnostic tool to assess fluid loading response or as a therapeutic maneuver pending fluid resuscitation.With the advantage of autotransfusion readily available,the Trendelenburg position is used for expected instantaneous effect on cardiovascular performance.
  Interventions: Diagnostic Test: Trendelenburg Maneuver
- dobutamine stress test (Experimental): Dobutamine is a selective beta 1 receptor agonist. It [<10 ug/(kg.min)] can effectively increase myocardial contractility.
  Interventions: Diagnostic Test: dobutamine stress test

INTERVENTIONS:
Diagnostic Test: Trendelenburg Maneuver — In the Trendelenburg position, the body is laid supine with the feet higher than the head by 15-30 degrees. The venous return increases in the trendelenburg position which in turn increases the stroke volume.
  Arms: Trendelenburg Maneuver
Diagnostic Test: dobutamine stress test — Dobutamine was infused intravenously at the initial dose of 2.5 ug/kg/min. Echocardiography was performed after 5-10 minutes of continuous infusion, and hemodynamic data were recorded.
  Arms: dobutamine stress test

SUMMARY:
Objective：

1. To evaluate the consistency of cardiac output measured by different hemodynamic monitoring methods in patients with VA-ECMO
2. To evaluate whether different hemodynamic monitoring methods can accurately detect the trend of cardiac output changes

DETAILED DESCRIPTION:
Venoarterial extracorporeal membrane oxygenation (VA-ECMO) has been used for profound cardiogenic shock to bridge to decision,ventricular assist devices,or transplant.Close monitoring of cardiac output, especially in patients before and after intervention (such as volume expansion, diuresis, vasoconstriction, vasodilation therapy), can help to adjust the treatment strategy. Hemodynamic monitoring in ECMO patients requires familiarity with the underlying pathophysiology and circulatory mechanics of extracorporeal flow.Limited to the actual clinical situation of patients, one or two hemodynamic monitoring methods may be accepted. Is there consistency between different hemodynamic monitoring results? And whether hemodynamic monitoring can accurately detect the changes of these parameters before and after intervention is an important issue in clinical practice. This study will provide important reference for VA-ECMO patients how to choose appropriate hemodynamic monitoring tools and how to interpret the results of hemodynamic monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. cardiac surgery
2. treatment with VA-ECMO
3. mechanical ventilation
4. hemodynamic monitoring according to patient's condition (PAC, Flotrac, echocardiography)

Exclusion Criteria:

1. age < 18
2. cardiac arrhythmia
3. moderate to severe aortic, mitral and tricuspid regurgitation
4. active hemorrhage
5. IABP
6. spontaneous triggering of the ventilator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Baseline Cardiac Output measurement | within1 minute at baseline position
  Cardiac Output measured at baseline position（ in a supine position with the head elevated to 15° for baseline measurements ）
Cardiac Output measurement afterTrendelenburg Maneuver | 1 minute after starting Trendelenburg Maneuver
  Cardiac Output measured after Trendelenburg Maneuver
Cardiac Output measurement after Dobutamine stress test | 5 minutes after dobutamine stress test
  Cardiac Output measured after dobutamine stress test

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, Doctor, Study Chair — Fudan University
Locations (1):
- Zhongshan hospital, Fudan university, Shanghai, China